CLINICAL TRIAL: NCT05107206
Title: Envi™-SR Randomized Controlled Trial for Endovascular Treatment of Ischemic Stroke
Acronym: ENVI RCT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was terminated due to management decision. Study was not terminated due to safety reasons.
Sponsor: NeuroVasc Technologies (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CL-001
Record Dates: First submitted 2021-10-21; First posted 2021-11-04 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Intervention Model Description: a prospective, multinational, randomized (adaptive), parallel group controlled, blinded, non-inferiority study.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Envi™-SR Thrombectomy Device (Experimental): Mechanical Thrombectomy using the Envi™-SR Thrombectomy Device
  Interventions: Device: Mechanical Thrombectomy using the Envi™-SR Thrombectomy device
- Solitaire or Trevo Revascularization Device (Active Comparator): Mechanical Thrombectomy using the Solitaire or Trevo Revascularization Device
  Interventions: Device: Mechanical Thrombectomy using the Solitaire or Trevo Revascularization Device

INTERVENTIONS:
Device: Mechanical Thrombectomy using the Envi™-SR Thrombectomy device — Clot removal using the Envi™-SR Thrombectomy device
  Arms: Envi™-SR Thrombectomy Device
Device: Mechanical Thrombectomy using the Solitaire or Trevo Revascularization Device — Clot removal using the Solitaire or Trevo Revascularization Device
  Arms: Solitaire or Trevo Revascularization Device

SUMMARY:
The study objective is to examine and compare clinical outcomes, as measured by Modified Rankin Scale (mRS) at 90 days (± 15 days) post treatment, and related performance characteristics of the Envi™-SR and concurrent parallel Control Devices currently cleared by the U.S. FDA for treatment of stroke.

DETAILED DESCRIPTION:
This study intends to evaluate a novel mechanical thrombectomy device to treat patients suffering from acute ischemic stroke through a prospective, randomized pivotal study to provide an assessment of the safety and non-inferiority of the device.

ELIGIBILITY:
Inclusion Criteria

1. Clinical signs consistent with acute ischemic stroke
2. Pre-stroke Modified Rankin Score ≤ 2
3. Age 18 years and no upper limit (patient must be 18 years old at time of consent).
4. NIHSS ≥ 6 at the time of randomization
5. Subject is able to start treatment (defined as time of arterial puncture) within 24 hours of stroke onset or last known well and within 90 minutes from last baseline CT/ MRI.
6. Imaging: For strokes in the anterior circulation the following imaging criteria should also be met:

   1. If stroke onset (as defined by the time the patient was last seen at baseline) is within 6 hours: Baseline ASPECTS ≥6 on non-contrast CT (NCCT) or DWI-MRI;
   2. If stroke onset is within 6-24 hours, advanced imaging with either CT perfusion or DWI-MRI is required. Baseline infarct volume must be ≤50cc for patients under 80 years old and ≤20cc for patients 80 years or older.
7. Location: Angiographic confirmation of an occlusion of an ICA (including T or L occlusions), M1 or M2 MCA, with eTICI flow of zero (0) - one (1).
8. Patients for whom IV t-PA is indicated are treated with IV t-PA without delay.
9. IV t-PA, if used, is initiated within three (3) hours of stroke onset (onset time is defined as the last time when the patient was witnessed to be at baseline), with investigator verification that the subject has received/is receiving the correct IV t-PA dose for the estimated weight.
10. Consent: The patient or the patient's legally authorized representative (LAR) has signed and dated an Informed Consent Form.
11. Will comply with protocol follow-up schedule.
12. Patient was ambulatory prior to stroke, i.e. able to walk without another person's assistance.

Exclusion Criteria

1. Life expectancy likely less than six (6) months.
2. Females who are pregnant or breastfeeding.
3. Known history of severe allergy (more than rash) to contrast medium that cannot be medically controlled.
4. Suspicion of renal failure (Renal failure as defined by a serum creatinine >3.0 mg/dL (264 μmol/L) or Glomerular Filtration Rate (eGFR) <30).
5. Severe, sustained hypertension (Systolic Blood Pressure >185 mmHg or Diastolic Blood Pressure >110 mmHg) NOTE: If the blood pressure can be successfully reduced and maintained at the acceptable level using medication the subject can be enrolled.
6. Currently participating in another interventional (drug, device, etc.) research project that may confound the results of this study.
7. Known hereditary or acquired hemorrhagic diathesis, coagulation factor deficiency. (A subject without history or suspicion of coagulopathy does not require INR or prothrombin time lab results to be available prior to enrollment.)
8. Known history of platelet count <100,000/μL.
9. Baseline blood glucose of <50mg/dL (2.78 mmol) or >400mg/dL (22.20 mmol).
10. Subjects with occlusions in multiple vascular territories (e.g., bilateral anterior circulation, or anterior/posterior circulation).
11. CT or MR evidence of hemorrhage.
12. Seizures at stroke onset.
13. Suspicion of aortic dissection.
14. Patients with known hypersensitivity to nickel-titanium.
15. Evidence of dissection in the extra or intracranial cerebral arteries.
16. Stenosis, or any occlusion, in a proximal vessel that requires treatment or prevents access to the site of occlusion.
17. Presumed septic embolus, suspicion of bacterial endocarditis, or other serious infection.
18. Suspected cerebral vasculitis based on medical history and CTA/Magnetic Resonance Angiogram (MRA).
19. Excessive vascular access tortuosity that will likely prevent endovascular access.
20. Baseline CT or Magnetic Resonance Imaging (MRI) showing intracranial tumor (except asymptomatic small meningiomas less than three (3) cm).
21. Significant mass effect with midline shift
22. Treatment with any cleared thrombectomy devices or other intra-arterial (neurovascular) therapies three months prior to use of treatment device
23. Unlikely to be available for 90-day (± 15 days) follow-up (e.g. no fixed home address, visitor from overseas).
24. Rapid neurological improvement prior to study enrollment suggesting resolution of signs/symptoms of stroke such as a decrease that leads to an NIHSS below the study cut-off of six (6).
25. Patient has suffered a hemorrhagic or ischemic stroke or TIA in at least the last three (3) months.
26. Patients with a pre-existing neurological or psychiatric disease that would confound the neurological or functional evaluations, mRS score at baseline must be ≤ 2. This excludes patients who are severely demented, require constant assistance in a nursing home type setting or who live at home but are not fully independent in activities of daily living (toileting, dressing, eating, cooking and preparing meals, etc.).
27. Known cancer with metastases.
28. Subject currently uses or has a recent history of illicit drug(s), which includes marijuana.
29. Recent past history (within three (3) months) or clinical presentation of intracranial hemorrhage (ICH), subarachnoid hemorrhage (SAH), ruptured arteriovenous malformation (AVM) or ruptured aneurysm.
30. The patient is in a coma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-06-23 (Actual); Primary Completion 2023-05-18 (Actual); Study Completion 2025-01-27 (Actual)

PRIMARY OUTCOMES:
Primary Effectiveness Endpoint: Proportion of subjects with good clinical outcome defined as Modified Rankin Score (mRS) of ≤2 | 90 days
  The proportion of subjects with good clinical outcome defined as Modified Rankin Score (mRS) of ≤2 as assessed by a blinded assessor at 90 days (± 15 days).
Primary Safety Endpoint: Device-related or procedure-related symptomatic intracranial hemorrhage (sICH) | 24 hours
  Device-related or procedure-related symptomatic intracranial hemorrhage (sICH) defined by the Heidelberg Bleeding Classification at 24 hours (-8/+12 hours) (as read by the Core Lab and adjudicated by Clinical Events Committee (CEC)).

CONTACTS AND LOCATIONS:
Overall Officials: Vitor Mendes-Pereira, MD, MSc, Principal Investigator — St Michael's Hospital and the University of Toronto; Raul G Nogueira, MD, Principal Investigator — University of Pittsburgh Medical Center
Locations (4):
- United States (4):
  - Providence Medical Foundation, Irvine, California
  - Baptist Health Research Institute, Jacksonville, Florida
  - Advocate Aurora Health, Downers Grove, Illinois
  - North Shore University Hospital, Manhasset, New York

IPD SHARING:
Plan to Share IPD: No